CLINICAL TRIAL: NCT03883815
Title: The Effect of Video Based Game Therapy on Activity Amount and Energy Consumption in Children With Cerebral Palsy
Brief Title: The Effect of Video-based Game Therapy on Treatment Intensity in Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Pınar Ciddi, lecturer assistant, doctor, Medipol University
Other Study IDs: 10840098-604.01.01-E.26936
Record Dates: First submitted 2019-03-10; First posted 2019-03-21 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; neurodevelopmental therapy; active video games; treatment intensity; energy consumption
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assesment treatment intensity: Assesment treatment intensity during neurodevelopmental therapy session and active video games therapy session
  Interventions: Other: Active Video Games Therapy

INTERVENTIONS:
Other: Active Video Games Therapy — Interventions were completed in 1-week periods, after 3 clinical visits. All individuals underwent both neurodevelopmental therapy and active video games therapy. Demographic data of individuals were recorded and muscle tone and gross motor functions were evaluated at the first visit. The games determined by the physiotherapist were explained and experienced by individuals. During the second visit, individuals played 4 games that were previously determined and experienced for about 45 minutes. On the last visit, individuals underwent neurodevelopmental therapy. During both treatment sessions, the accelerometer was fitted on a flexible belt by attaching it to the dominant wrist. Individuals were instructed not to remove the device during both treatment sessions.
  One session individuals treated with exercises which weight transfer and postural reactions were facilitated.
  Other session they played Nintendo Wii games in accordance with their current level and skills.
  Other Names: Neurodevelopmental therapy

SUMMARY:
In a recent review by Kolobe et al., It was reported that there was no study investigating the effects of treatment intensity on upper or lower extremity function in children with traumatic brain injury and cerebral palsy. In other words, any study in this review reported no studies on the amount of effort or the number of repetitions at high or low intensity.

This indicates a clear gap in the literature related to density, which is a dosage variable for cerebral palsy.

It is difficult to determine and increase density without having strong, practical methods to measure density during rehabilitation.

Therefore, there is a clear need for alternative measurements to measure density.

As the alternative measurements, the number of repetitions, the duration of active time during the sessions are used.

Energy consumption seen as a useful tool for evaluating functional capacity may also reflect activity intensity by measuring the intensity of activity during the session.

Because the ability to perform an activity when interpreted; It is considered as an indicator of fatigue and endurance.

Children with cerebral palsy have decreased selective muscle control, abnormal muscle tone, imbalance between agonist and antagonist muscles, and abnormalities in balance due to inadequate balance reactions.

Due to all these reasons, cerebral palsy in children has been shown to have higher energy consumption during physical activities such as walking compared to healthy children.

Children with cerebral palsy usually have difficulty in regular participation in treatment and adaptation to traditional home exercise programs. Active video games are recommended for use in addition to neurodevelopmental therapy and, in particular, for home use, because of the potential for increasing treatment dosage.

Researchers focus on evidence in terms of exercise games, Some games on the market (Wii Sports tennis and boxing and Dance Dance Revolution) have achieved that the physical activity measured by the metabolic equivalent, which is necessary to perform the tasks in individuals with cerebral palsy, is associated with the level of moderate severity.

In this study, it is aimed to compare the treatment intensity, performance and balance parameters of the patients with cerebral palsy in a planned neurodevelopmental treatment session and active video games.

In this study, the effects of clinical type, age and functional level on treatment intensity, performance and balance parameters during these sessions will be investigated.

Hypothesis of the study In line with the needs of children with cerebral palsy, there is a difference in terms of treatment intensity, performance and balance parameters between a planned neurodevelopmental treatment session and active video games.

ELIGIBILITY:
Inclusion Criteria:

1. Having a diagnosis of cerebral palsy by a qualified physician, between the ages of 6-18 and continuing ambulations,
2. Functional to Gross Motor Function Classification System be between levels I-III,
3. To be cooperative during the evaluation and treatment sessions,
4. Individuals do not have a history of genetic and / or neurological disease other than cerebral palsy,
5. In terms of the movements of the upper extremities; Should be able to shoulder flexion up to 90 degrees, have enough functional hand ability to grasp the Nintendo Wii control, actively flex elbow and extension within the functional limits, lack of spasticity of the upper extremity muscles which may interfere with all these movements,
6. To be able to play the game with sufficient balance to be able to stand,
7. Have not played Nintendo Wii before,
8. There is no defect in the visual functions except breakage defect

Exclusion Criteria:

1. Passing muscle-tendon and bone operation less than 6 months ago,
2. have been exposed to any pharmacological agent to inhibit spasticity within 6 months,
3. have cognitive / mental problems that will interfere with communication with him / she will not understand working instructions,
4. Difficulty in visual functions except for fracture failure,
5. A history of genetic and / or neurological disease other than cerebral palsy,
6. The patient was negatively affected by physical activity and was diagnosed as having epileptic seizures.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Individuals with a diagnosis of Cerebral Palsy who had been undergoing physiotherapy for 2 days a week between the ages of 6 and 18 were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-08-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
energy consumption | 45 minutes
  data on energy consumption during sessions obtained as a result of accelerometer device (in Metabolic Equivalence)

SECONDARY OUTCOMES:
number of activities | 45 minutes
  data on acitivity numbers during sessions obtained as a result of accelerometer device (in counts)
active time during session | 45 minutes
  data on active time during sessions obtained as a result of accelerometer device (in minutes)

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Istanbul, Eyalet/Yerleşke, Turkey (Türkiye)